CLINICAL TRIAL: NCT02482740
Title: An Open, Randomized, Multi-center, Phase 2 Trial of Tamoxifen and Letrozole in Recurrent and Persistent Squamous Cell Carcinoma of the Cervix: the Efficacy and New Biomarkers
Brief Title: A Trial of Tamoxifen and Letrozole in Recurrent and Persistent Squamous Cell Carcinoma of the Cervix
Acronym: TGOG1005
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Collaborators: Chang Gung Memorial Hospital (Other); Chung Shan Medical University (Other); China Medical University Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Kaohsiung Veterans General Hospital. (Other); Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Tang Yuan Chu, The Chief of Department of Obstetrics and Gynecology, Buddhist Tzu Chi General Hospital, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TGOG1005
Record Dates: First submitted 2015-05-12; First posted 2015-06-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Uterine Cervical Neoplasms; antiestrogens
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Letrozole; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tamoxifen (Experimental): tamoxifen 20 mg given everyday for 12 months
  Interventions: Drug: tamoxifen
- letrozole (Active Comparator): letrozole 2.5 mg given everyday for 12 months
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — letrozole 2.5 mg qd was given for 12 months or till disease progress
  Other Names: Femara
  Arms: letrozole
Drug: tamoxifen — tamoxifen was given 20 mg qd for 12 months or till disease progress
  Other Names: Nolvadex
  Arms: tamoxifen

SUMMARY:
The investigators design a phase 2, open labeled, randomized trial of Tamoxifen (20 mg/day) and Letrozole (2.5 mg) in treatment of squamous carcinoma of the cervix. Forty four patients with recurrent or persistent disease will be recruited, randomized, treated and followed three-monthly for 12 months. The primary end point is the treatment response rates. Secondary end points include survivals, ECOG performance status, quality of life and efficacy of biomarkers in predicting the responses. Candidate biomarkers including ER, PR, GPER and HPV genotype in paraffin cancer tissues as well as methylated genes in the blood will be studied in relation to the therapeutic outcomes.

DETAILED DESCRIPTION:
Although human papillomavirus (HPV) is a necessary cause of cervical cancer, HPV infection itself is inefficient and insufficient to cause cancer. New evidences have suggested endogenous and exogenous sex hormones confer risk of developing cervical cancer. In unscreened populations, incidence of cervical cancer starts after menarche and constantly increases before menopause, after then the incidence is flattening and declines [21]. Indeed, after menopause, newly incident CIN3 is seldom detected[22]. Large-scale epidemiological studies also showed high number of full-term pregnancy[23] (rather than abortion) and long-term use of hormonal contraceptives[24] to be independent risk factors of cervical cancer. These evidences pointed to female sex hormones to be another culprit of cervical cancer.

The role of estrogen and ERα on HPV-induced cervical carcinogenesis is best demonstrated by the pK14-HPV E6/E7transgenic mice which, without estrogen exposure, develop benign skin tumors only. However, when these mice are treated with exogenous estradiol at physiological level, they develop cervical cancers in nearly 100% efficiency[25-28]. These cervical neoplasia recapitulate characteristics of human cervical cancer in all aspects: originated from the squamous-columnar junction, with early lesions of atypical squamous metaplasia, CIN and to invasive squamous cell carcinoma [29]. Most importantly, removal of exogenous estrogen or castration of these mice led to diminish of progression and partial regression of pre-existing neoplasia[30].

The investigators design an open, randomized, multi-center trial of tamoxifen and letrozole in treatment of recurrent or persistent squamous cell carcinoma of the cervix. Patients with recurrent or persistent SCC of cervix who are not amenable for further cytotoxic treatment will be randomized by block and by participating center to one of the two arms. The block size will be two . Medication will be given orally in daily dose of tamoxifen (Nolvadex) 20 mg, letrozole (Femara) 2.5 mg until disease progression or until the end of the study.

Primary end point of the study is the response rate (complete response and partial response rates) for tamoxifen and letrozole arms. Secondary end points include progression-free survival (PFS) and overall survival (OS) compared to the historical results, ECOG Performance Status, quality of life and outcome predictors (biomarkers and clinical characteristics) of responsiveness and survival. The experienced survival data of the participating center will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. With a histology proven primary squamous cell carcinoma of the cervix prior to the treatment failure
2. Must sign and date informed consent.
3. With age between 30 and 85
4. With tissue blocks of the recurrent cancer lesion or primary cancer lesion available for the study.
5. With a treatment-free interval of at least 4 weeks.
6. With currently (within 1 month) measurable (by CT) tumor of at least 2 cm in one diameter (at least twice the scan slice thickness), AND elevated SCC level over 2 folds of the institutional upper limit of normal (ULN),
7. With a ECOG performance status score of 0 to 2,
8. With adequate hematologic function (ANC≧500/uL and platelets≧50,000/uL),
9. With adequate renal function (serum creatinine≦2.0 mg/dL; if higher, then creatinine clearance≧40 mL/min was required),
10. With adequate hepatic function (ALT/AST ≦3.0 folds of ULN

Exclusion Criteria:

1. With histology type other than SCC
2. Had liver, brain metastasis or malignant ascites
3. Those having multiple metastasis (more than one metastasis lesion)
4. Whose cancer had been treated for more than three therapeutic courses [including 1 primary therapy (Operation+ CCRT is considered 1 primary therapy) and 2 secondary therapies] courses.
5. Who have received any investigational drugs within 30 days prior to enrollment
6. Who were pregnant or lactating
7. Who are taking selective serotonin receptor inhibitors (SSRI) (eg. Prozac, Celexa, Lexapro, Lubox, Paxi, Zoloft, etc.)
8. With pulmonary embolism or other veneous embolism
9. With uncontrolled medical conditions such as cardiac disease, cirrhosis of liver, active on chronic hepatitis, diabetes mellitus, autoimmune disease.
10. With current or prior therapy (less than 3 months ) of selective estrogen receptor modulators (SERMs) (tamoxifen, raloxifen, fulvestrant, etc.), or aromatase inhibitors (eg. Letrozole, Anastrozole, Exemestane, Vorozole, Formestane, Fadrozole, etc.)
11. Currently taking Warfarin or Rivaroxaben .
12. With history of malignant disease, except those had been disease-free for at least 5 years.
13. Patient who had allergy history to Tamoxifen or Letrozole

Ages: 30 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The response rate | one year
  The guideline for the Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1) will be followed. Target tumor will be identified and followed by CT scan. Other efficacy parameters are tumor markers (SCC), and pelvic examination and physical examination findings.

SECONDARY OUTCOMES:
Progression-free survival | one year
  Progression-free survival (PFS) comparing to the historical results
Quality of life | one year
  The European Organization for Research and Treatment of Cancer (EORTC) Quality-of-Life questionnaire cervical cancer module: EORTC QLQ-CX24 and C30 will be evaluated for every patient at every visit during study period.
ECOG Performance Status | one year
  ECOG Performance status will be evaluated every visit during study period
Overall survival | one year
  overall survival (OS) comparing to the historical results

CONTACTS AND LOCATIONS:
Overall Officials: Tang Yuan Chu, PhD, Principal Investigator — Department of Obstetrics and Gynecology, Buddhist Tzu Chi General Hospital, 707, Section 3, Chung Yang Road, Hualien 970, Taiwan (R.O.C.)
Locations (7):
- Taiwan (7):
  - Dept. of Obstetrics and Gynecology, Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, No 123, Dapi Rd, Niaosong Dist
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, No.100, Ziyou 1st Rd., Sanmin Dist.
  - Chung Shan Medical University Hospital, Taichung, No.110,sec. 1,Jianguo NRd.,South Dist.
  - National Cheng Kung University Hospital, Tainan, No.138, Shengli Rd., North Dist.
  - China Medical University Hospital, Taichung, No.2, Yude Rd., North Dist.,
  - Kaohsiung Veterans General Hospital, Kaohsiung City, No.386, Dazhong 1st Rd., Zuoying Dist.
  - Department of OB/GYN, Linkou Chang Geng Memorial Hospital, Taoyuan District, Taoyuan

REFERENCES:
- [Background] Plummer M, Peto J, Franceschi S; International Collaboration of Epidemiological Studies of Cervical Cancer. Time since first sexual intercourse and the risk of cervical cancer. Int J Cancer. 2012 Jun 1;130(11):2638-44. doi: 10.1002/ijc.26250. Epub 2011 Aug 12. PMID 21702036
- [Background] Rodriguez AC, Schiffman M, Herrero R, Hildesheim A, Bratti C, Sherman ME, Solomon D, Guillen D, Alfaro M, Morales J, Hutchinson M, Katki H, Cheung L, Wacholder S, Burk RD. Longitudinal study of human papillomavirus persistence and cervical intraepithelial neoplasia grade 2/3: critical role of duration of infection. J Natl Cancer Inst. 2010 Mar 3;102(5):315-24. doi: 10.1093/jnci/djq001. Epub 2010 Feb 15. PMID 20157096
- [Background] International Collaboration of Epidemiological Studies of Cervical Cancer. Cervical carcinoma and reproductive factors: collaborative reanalysis of individual data on 16,563 women with cervical carcinoma and 33,542 women without cervical carcinoma from 25 epidemiological studies. Int J Cancer. 2006 Sep 1;119(5):1108-24. doi: 10.1002/ijc.21953. PMID 16570271
- [Background] International Collaboration of Epidemiological Studies of Cervical Cancer; Appleby P, Beral V, Berrington de Gonzalez A, Colin D, Franceschi S, Goodhill A, Green J, Peto J, Plummer M, Sweetland S. Cervical cancer and hormonal contraceptives: collaborative reanalysis of individual data for 16,573 women with cervical cancer and 35,509 women without cervical cancer from 24 epidemiological studies. Lancet. 2007 Nov 10;370(9599):1609-21. doi: 10.1016/S0140-6736(07)61684-5. PMID 17993361
- [Background] Riley RR, Duensing S, Brake T, Munger K, Lambert PF, Arbeit JM. Dissection of human papillomavirus E6 and E7 function in transgenic mouse models of cervical carcinogenesis. Cancer Res. 2003 Aug 15;63(16):4862-71. PMID 12941807
- [Background] Shai A, Brake T, Somoza C, Lambert PF. The human papillomavirus E6 oncogene dysregulates the cell cycle and contributes to cervical carcinogenesis through two independent activities. Cancer Res. 2007 Feb 15;67(4):1626-35. doi: 10.1158/0008-5472.CAN-06-3344. PMID 17308103
- [Background] Arbeit JM, Howley PM, Hanahan D. Chronic estrogen-induced cervical and vaginal squamous carcinogenesis in human papillomavirus type 16 transgenic mice. Proc Natl Acad Sci U S A. 1996 Apr 2;93(7):2930-5. doi: 10.1073/pnas.93.7.2930. PMID 8610145
- [Background] Elson DA, Riley RR, Lacey A, Thordarson G, Talamantes FJ, Arbeit JM. Sensitivity of the cervical transformation zone to estrogen-induced squamous carcinogenesis. Cancer Res. 2000 Mar 1;60(5):1267-75. PMID 10728686
- [Background] Brake T, Connor JP, Petereit DG, Lambert PF. Comparative analysis of cervical cancer in women and in a human papillomavirus-transgenic mouse model: identification of minichromosome maintenance protein 7 as an informative biomarker for human cervical cancer. Cancer Res. 2003 Dec 1;63(23):8173-80. PMID 14678972
- [Background] Brake T, Lambert PF. Estrogen contributes to the onset, persistence, and malignant progression of cervical cancer in a human papillomavirus-transgenic mouse model. Proc Natl Acad Sci U S A. 2005 Feb 15;102(7):2490-5. doi: 10.1073/pnas.0409883102. Epub 2005 Feb 7. PMID 15699322